CLINICAL TRIAL: NCT04995016
Title: A Single-center, Non-randomized Controlled, Single-arm, Phase II Clinical Trial of Pembrolizumab and Axitinib as Neoadjuvant Therapy for Locally Advanced Non-metastatic Clear Cell Renal Cell Carcinoma
Brief Title: Pembrolizumab and Axitinib as Neoadjuvant Therapy for Locally Advanced Non-metastatic Clear Cell Renal Cell Carcinoma
Acronym: PANDORA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANDORA 001
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma
Keywords: Pembrolizumab; Axitinib; Neoadjuvant
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pembrolizumab; Axitinib

STUDY DESIGN:
Intervention Model Description: simon's two stage design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Locally Advanced Non-metastatic Clear Cell Renal Cell Carcinoma (Experimental): Neoadjuvant pembrolizumab plus axitinib
  Interventions: Drug: Pembrolizumab; Drug: Axitinib

INTERVENTIONS:
Drug: Pembrolizumab — PD-1 inhibitor，Pembrolizumab 200mg IV, every 3 weeks.
  Other Names: Keytruda
Drug: Axitinib — Tyrosine kinase inhibitor，licensed for use in treatment of renal cell carcinoma. Oral treatment Axitinib given 5 mg PO BID.
  Other Names: Inlyta

SUMMARY:
This is a single-arm phase II clinical trial to evaluate the initial efficacy and safety of pembrolizumab combined with axitinib as neoadjuvant therapy for locally advanced non-metastatic clear cell renal cell carcinoma.

DETAILED DESCRIPTION:
This study is design to prospectively investigate the safety and efficacy of pembrolizumab combined with axitinib in downsizing tumors in patients with nonmetastatic biopsy-proven clear cell renal cell carcinoma. This is a single-institution, single-arm phase 2 clinical trial. Patients will receive axitinib 5 mg bid on days 1-21 combined with pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatments repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.Patients then will receive partial or radical nephrectomy after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a renal mass consistent with a clinical stage >= T3Nx or TanyN+ or deemed unresectable by surgeon
* Renal cell carcinoma with clear cell component on pre-treatment biopsy of the primary tumor
* The participant (or legally acceptable representative if applicable) provides written informed consent and the willingness and ability to comply with all aspects of the protocol
* Have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Agree to collect tumor tissue, blood and other specimens required by this study and apply them to relevant studies
* Important organs and bone marrow functions meet the following requirements: absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet (PLT) ≥100×10^9/L, hemoglobin (HGB) ≥9g/dL;Liver function: serum total bilirubin (TBIL) ≤1.5 times normal upper limit (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 times ULN, serum albumin (ALB) ≥ 2.8g /dL. Renal function: serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥40 mL/min
* Cardiac function met the following conditions: baseline electrocardiogram (ECG) had no evidence of PR prolongation or AV block
* All females must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [beta-hCG]) at the screening visit and the baseline visit. A pregnancy test needs to be performed within 72 hours of the first dose of study drug. Women of childbearing potential (WOCBP) must agree to use a highly effective method of contraception for the entire study period and for 120 days after study discontinuation
* Male subjects who are partners of women of childbearing potential must use a condom and their female partners of childbearing potential must use a highly effective method of contraception beginning at least 1 menstrual cycle prior to starting study drugs, throughout the entire study period, and for 120 days after the last dose of study drug, unless the male subjects are totally sexually abstinent or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile

Exclusion Criteria:

* Subject has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents
* Subject is currently participating or has participated in a study of an investigational agent or using an investigational device within 30 days of the first dose of study treatment
* Subject is expected to require any other form of systemic or localized antineoplastic therapy while on study
* Subject is on any systemic steroid therapy, within one week before the planned date for first dose of study treatment.
* Subject is on any other form of immunosuppressive medication
* Unable to swallow and retain orally administered medication
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other -Gastrointestinal conditions with increased risk of perforation; history of abdominal fistula, GI perforation, or intra-abdominal abscess within 4 weeks before beginning study treatment
* Known history of HIV infection or a known history of or is positive for Hepatitis B or Hepatitis C
* Presence of active infection requiring systemic therapy
* Corrected QT interval duration prolongation
* History of any one or more of the following cardiac conditions within the past 6 months: Cardiac angioplasty or stenting; Myocardial infarction; Unstable angina; --History of Class III or IV congestive heart failure according to New York Heart Association classification
* History of cerebrovascular accident within the past 6 months
* Poorly controlled hypertension
* History of untreated deep venous thrombosis
* Presence of any non-healing wound, fracture, or ulcer, or presence of symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Has taken any prohibited medications that are listed in the protocol within 14 days of the first dose of study treatment
* Subject has received or will receive a live vaccine within 30 days before the first administration of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2022-08-20 (Estimated); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) | 12 weeks
  The residual tumor cells (% RVT) were calculated according to immune related pathologic response criteria (irPRC), MPR is defined as %RVT<10%

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) | 12 weeks
  The residual tumor cells (% RVT) were calculated according to immune related pathologic response criteria (irPRC), pCR is defined as %RVT<0%
Objective response rate (ORR) | 12 weeks
  Rate of patients achieving a complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and immune-related response criteria (IRC)
Disease-free survival(DFS) | Up to 24 months
  DFS is defined as the time from treatment to recurrence of tumor or death
Overall survival(OS) | Up to 24 months
  OS is defined as the time from treatment to death
Incidence of treatment-related adverse events(AEs) | Up to 24 months
  To be assessed by CTCAE v5.0

OTHER OUTCOMES:
Biomarker analysis | Up to 24 months
  Paired t-test or Wilcoxon singed-rank test will be used to compare the biomarkers change before, during, and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bin HUO, MD, Principal Investigator — Tianjin Medical University Second Hospital; Gang LI, MD, Principal Investigator — Tianjin Medical University Second Hospital; Haitao WANG, Professor, Study Director — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No